CLINICAL TRIAL: NCT06220175
Title: Pharynx Analgesia Before Upper Gastrointestinal Endoscopy: a Prospective, Randomized Comparative Trial
Brief Title: Pharynx Analgesia Before Upper Gastrointestinal Endoscopy
Acronym: PHRASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Associate Professor of Gastroenterology, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRASE
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Upper Gastrointestinal Endoscopy
MeSH Terms: interventions — Strepsils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strepsils Intensiv Arm + Xilocaine Spray (Experimental): Patient will take one pill of Strepsils Intensiv containing 8.75mg flurbiprofen 10 to 15 minutes before endoscopy.
  The patient will have pharyngeal topical xilocaine spray before upper GI endoscopy, 5 puffs in two applications immediately before examination.
  Interventions: Drug: Strepsils Intensiv plus Xilocaine spray Arm
- Xilocaine Spray Arm (Active Comparator): The patient will have pharyngeal topical xilocaine spray before upper GI endoscopy, 5 puffs in two applications immediately before examination.
  Interventions: Drug: Xilocaine Spray Arm

INTERVENTIONS:
Drug: Strepsils Intensiv plus Xilocaine spray Arm — After Stepsils Intensiv ingestion, upper GI endoscopy will be performed with a standard diameter tube, with SpO2 non invasive monitoring.
  Other Names: Strepsils + Xilocaine Spray
  Arms: Strepsils Intensiv Arm + Xilocaine Spray
Drug: Xilocaine Spray Arm — After Xilocaine Spray pharyngeal topical anestesia, upper GI endoscopy will be performed with a standard diameter tube, with SpO2 non invasive monitoring.
  Other Names: Xilocaine
  Arms: Xilocaine Spray Arm

SUMMARY:
This is a comparative study on patient and endoscopist experience during upper gastrointestinal endoscopy with NSAIDs (flurbiprofen) topical analgesia plus xilocaine spray topical anesthesia of the pharynx versus xilocaine spray topical anesthesia of the pharynx alone, before procedure.

DETAILED DESCRIPTION:
Upper gastrointestinal endoscopy may be done with topical anesthesia of the pharynx with xilocaine spray, with conscious sedation with midazolam or with general anesthesia with propofol. In Romania, the endoscopist may only offer topical pharyngeal anesthesia, any other sedation or anesthesia needs the presence of an anesthesiologist on premises.

Xilocaine spray improves the gag reflux and the satisfaction score of the patient as well as the ease of insertion and the satisfaction score of the endoscopist.

A study published in 2010 has compared the tolerance of upper GI endoscopy in patients in which the topical anesthesia of the pharynx has been done using Strepsils Plus with xilocaine versus xilocaine spray. The group of patients with Strepsils Plus had a significantly lower tolerance, lower anesthesia score, a higher gag score and a higher disconfort score versus patients in group with xilocaine spray.

Nevertheless, topical pharyngeal anesthesia with benzocaine spray and in much lesser degree with xilocaine spray may lead to a very rare adverse reaction, namely methemoglobinemia. That is why, an safer alternative to xilocaine spray would be desirable at this moment.

Question at which the research protocol is trying to answer The investigators intent to evaluate whether a topical pharyngeal anti inflammatory molecule, a non steroidal anti inflammatory drug (NSAID), that is Strepsils Intensive with honey and lemon which contains flurbiprofen 8.75mg before upper GI endoscopy plus xilocaine spray improves the satisfaction score of the patient as compared to standard xilocaine spray alone.

Hypothesis A topical NSAID will improve the satisfaction score of the patient during upper GI endoscopy, when added to xilocaine spray.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication of upper gastrointestinal endoscopy with topical pharyngeal anesthesia with xilocaine spray
* Age above 18 years
* Informed consent

Exclusion Criteria:

* Allergy to xilocaine and/or flurbiprofen
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction score | 24 hours
  Evaluation on visual score 0 - 10 (0 - minimum, 10 - maximum)

SECONDARY OUTCOMES:
Patient discomfort score | 24 hours
  Evaluation on visual score 0 - 10 (0 - minimum, 10 - maximum)
Patient pain score | 24 hours
  Evaluation on visual score 0 - 10 (0 - minimum, 10 - maximum)
Patient gag score | 24 hours
  Evaluation on visual score 0 - 10 (0 - minimum, 10 - maximum), by the endoscopist
Endoscopist satisfaction score | 24 hours
  Evaluation on visual score 0 - 10 (0 - minimum, 10 - maximum)

CONTACTS AND LOCATIONS:
Locations (1):
- "Agrippa Ionescu" Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amornyotin S, Srikureja W, Chalayonnavin W, Kongphlay S, Chatchawankitkul S. Topical viscous lidocaine solution versus lidocaine spray for pharyngeal anesthesia in unsedated esophagogastroduodenoscopy. Endoscopy. 2009 Jul;41(7):581-6. doi: 10.1055/s-0029-1214865. Epub 2009 Jul 8. PMID 19588284
- [Background] Chan CK, Fok KL, Poon CM. Flavored anesthetic lozenge versus Xylocaine spray used as topical pharyngeal anesthesia for unsedated esophagogastroduodenoscopy: a randomized placebo-controlled trial. Surg Endosc. 2010 Apr;24(4):897-901. doi: 10.1007/s00464-009-0687-9. PMID 19730942
- [Background] Mahawongkajit P, Talalak N, Soonthornkes N. Comparison of Lidocaine Spray and Lidocaine Ice Popsicle in Patients Undergoing Unsedated Esophagogastroduodenoscopy: A Single Center Prospective Randomized Controlled Trial. Clin Exp Gastroenterol. 2021 May 25;14:209-216. doi: 10.2147/CEG.S301163. eCollection 2021. PMID 34079324